CLINICAL TRIAL: NCT02218918
Title: Phase 0 Study of Comparison Between Ground Walk Training and Treadmill Walk Training in COPD Patients
Brief Title: Comparison of Supervised Ground Walk Training and Treadmill Walk Training in COPD Patients
Acronym: GWT/TWT
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: PSG Hospitals (Other)
Responsible Party: Principal Investigator, Baskaran Chandrasekaran, Senior Physiotherapist, PSG Hospitals
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: PSG01Rehab
Record Dates: First submitted 2014-08-11; First posted 2014-08-18 (Estimated); Last update posted 2017-10-20 (Actual); Status verified 2017-10

CONDITIONS: Chronic Obstructive Pulmonary Disease (COPD)
Keywords: Ground walk; treadmill walk; Functional walk capacity; COPD; Quality of Life
MeSH Terms: conditions — Pulmonary Disease, Chronic Obstructive

STUDY DESIGN:
Intervention Model Description: Treadmill training vs ground walk training
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Supervised Treadmill Walk Training (Active Comparator): Based on 6 minute walk distance, treadmill speed initiated and progression on basis new 6 minute walk distance every 2 weeks
  Interventions: Behavioral: Supervised Treadmill Walk training
- Supervised Ground walk training (Experimental): Ground walk training progressed on the basis of 6 minute walk distance (70 - 90%), Weekly 3 days and for 6 weeks
  Interventions: Behavioral: Ground walk training

INTERVENTIONS:
Behavioral: Ground walk training — 3 times a week and 6 weeks
  Arms: Supervised Ground walk training
Behavioral: Supervised Treadmill Walk training — 3 times a week and 6 weeks
  Arms: Supervised Treadmill Walk Training

SUMMARY:
Pulmonary Rehabilitation became a vital part of management in COPD patients in form of activity modification, dietary and pharmacological optimisation. But access to traditional supervised aerobic (treadmill) walking is debatable fact due to economical and staffing expertise in developing countries like India. The investigators designed a randomised controlled trial to evaluate the effectiveness of ground based walking over traditional treadmill walking in improving quality of life in COPD patients.

DETAILED DESCRIPTION:
Background: COPD is increasing mortality and morbidity globally. Pulmonary rehabilitation is a promising management in COPD management. Exercise training in form of aerobic (walking, cycling) and strength training is an important part of pulmonary rehabilitation. However access to traditional supervised exercise programs is questionable debate even in developed western countries. Unsupervised ground walk programs are often told by physicians but not properly prescribed.

Objective: To assess whether ground or treadmill walk is better in improving functional capacity and quality of life in COPD patients Design: Randomised controlled trial Procedure: Two arms 1) supervised ground walk training 2) supervised treadmill walk training. The intensity and progression of walk is based on 6 minute walk test. Quality of life will be gauged through Chronic respiratory questionnaire and functional capacity through 6 minute walk test.

Statistical analysis: Descriptive analysis for characterisation. Normality though Kolmogorov and Variables will be compared through paired and unpaired student t tests

ELIGIBILITY:
Inclusion Criteria:

* stable COPD
* Stage II - IV
* Both genders

Exclusion Criteria:

* Cardiovascular diseases uncompensated
* uncompensated pleural diseases
* uncompensated liver diseases
* Recent surgeries less than 3 weeks
* malignancy receiving chemo and radiotherapy
* Recent exacerbations less than 3 months

Ages: 40 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Actual)
Dates: Start 2014-07 (Actual); Primary Completion 2016-08 (Actual); Study Completion 2016-10 (Actual)

PRIMARY OUTCOMES:
Functional Capacity (6 MINUTE WALK TEST) | Baseline, 6 weeks
  6 minute walk test according to standardisation of ATS
Quality of Life (Chronic Respiratory Questionnaire) | Baseline, 6 weeks
  CRQ - interviewer based

CONTACTS AND LOCATIONS:
Overall Officials: Baskaran Chandrasekaran, MPTh, Principal Investigator — Senior Physiotherapist
Locations (1):
- PSG Hospitals, Coimbatore, Tamil Nadu, India